CLINICAL TRIAL: NCT02639416
Title: Hypoallergenic and Anti-inflammatory Feeds to Treat Intestinal Inflammation in Malawian Children With Severe Acute Malnutrition: A Pilot Randomized Controlled Clinical Trial (SAM)
Brief Title: Hypoallergenic and Anti-inflammatory Feeds in Malawian Children With Severe Acute Malnutrition (SAM)
Acronym: SAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: University of Toronto (Other); Kamuzu University of Health Sciences (Other); Queen Elizabeth Central Hospital, Blantyre, Malawi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15.048
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Severe Malnutrition; Enteritis
Keywords: severe acute malnutrition; polymeric therapeutic formula; elemental therapeutic formula
MeSH Terms: conditions — Malnutrition; Enteritis; Severe Acute Malnutrition | interventions — Food, Formulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard management (Active Comparator): Standard management consists of F-100 and/or ready-to-use therapeutic food (RUTF) according to usual practice for 14 days
  Interventions: Other: Standard management
- Polymeric formula (Experimental): Exclusive polymeric formula supplemented with micronutrients in equivalent volume to F-100 for 14 days
  Interventions: Dietary Supplement: Polymeric formula
- Elemental formula (Experimental): Exclusive elemental formula supplemented with micronutrients in equivalent volume to F-100 for 14 days
  Interventions: Dietary Supplement: Elemental formula

INTERVENTIONS:
Dietary Supplement: Polymeric formula — Polymeric formulae are recommended in the management of inflammatory bowel disease in children
  Arms: Polymeric formula
Dietary Supplement: Elemental formula — Elemental formulae are recommended in cow's milk and other food intolerances in children.
  Arms: Elemental formula
Other: Standard management — Standard management with F-100 and/or RUTF
  Arms: Standard management

SUMMARY:
Children with complicated severe acute malnutrition (SAM), such as inability to take adequate feeds, infection and diarrhoea, require in-patient management. Despite following a well-established World Health Organisation (WHO) protocol, outcomes are poor. Case fatality often exceeds 20%. Amongst survivors discharged home, many subsequently die, have long-term poor growth or recurrence of SAM.

It has long been recognized that children with SAM have intestinal inflammation and that this persists despite management according to WHO guidelines. The inflammation is thought to result from increased exposure to microbial pathogens in the gut in areas with poor sanitation. The damaged lining of the intestine impairs food digestion and absorption, likely allows gut bacteria to enter the blood stream to cause sepsis and also exposes the gut immune cells to microbial and food antigens causing the inflammation to persist. Failure to treat the intestinal inflammation is likely to contribute to the poor response to treatment and poor long-term outcomes in many children with SAM.

The intestinal inflammation seen in SAM is very similar to that which occurs in food intolerance (e.g. intolerance to cow's milk protein) and inflammatory bowel disease. In these conditions, the inflammation is treated very effectively with hypoallergenic ("elemental") and anti-inflammatory ("polymeric") formulas. These are nutritionally complete feeds that have a similar composition to the feeds used for nutritional rehabilitation in SAM.

We aim to undertake a pilot study to see if an elemental and/or polymeric formula are tolerated by children with SAM and help to reduce intestinal inflammation. We also aim to learn more about the intestinal inflammation in general that occurs in SAM by observing carefully the effect of these specific formulae and to do in-depth metabolic analyses.

DETAILED DESCRIPTION:
We will study children admitted to the Moyo ward at the Queen Elizabeth Central Hospital, Blantyre, Malawi with complicated SAM. Following informed consent, children will be recruited once they have completed the initial stabilisation phase of management and enter the transition phase to nutritional rehabilitation. They will be randomly allocated to one of 3 arms, either 1) standard feeds (F-100 and/or ready-to-use therapeutic feeds), 2) a polymeric therapeutic formula or 3) an elemental therapeutic formula. The alternative feeds will be supplemented with micronutrients to be equivalent in composition to F-100. All children will remain admitted to the ward for 2 weeks and receive exclusively the allocated formula. All other aspects of the management of SAM will follow current practice based on WHO guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-23 months
* SAM diagnosed according to WHO criteria: (Weight-for-height z score <-3 and/or mid-upper arm circumference <11.5 cms and/or nutritional oedema)
* Admitted to hospital because of SAM with medical complications or fails an appetite test
* Completed stabilization phase and entering the second phase in refeeding; the transition Phase
* Willing to stay on the ward for 2 weeks after the stabilization phase (travel expenses will be provided)

Exclusion Criteria:

* Specific cause of malnutrition (e.g. cerebral palsy, other organ disease)
* Sibling admitted with SAM at the same time
* Unwilling to stay on ward for at least 2 weeks
* Declined to give consent
* Participating in another study

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-01-11 (Actual)

PRIMARY OUTCOMES:
Change in faecal calprotectin | 14 days
  Validated marker of intestinal inflammation

SECONDARY OUTCOMES:
Days with diarrhoea | 1-14 days
  number of days with 3 or more loose/watery stools
Weight gain | 1-14 days
  change in weight in g/kg/day
Episodes of sepsis | 1-14 days
  Clinical diagnosis
Death | 1-14 days
  number of children who die

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Allen, MD, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Moyo ward, Department of Paediatrics, Queen Elizabeth Central Hospital, Blantyre, Southern Region, Malawi

IPD SHARING:
Plan to Share IPD: Yes